CLINICAL TRIAL: NCT01740960
Title: Safety and Tolerability of Oral Namisol®, a Tablet Containing Delta-9-Tetrahydrocannabinol, in Elderly Subjects: A Randomized Controlled Trial
Brief Title: Safety and Tolerability of Namisol in the Elderly
Acronym: THC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GER001-02-03; 2012-001841-42 (EudraCT Number)
Record Dates: First submitted 2012-11-15; First posted 2012-12-04 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2012-07

CONDITIONS: Drug Safety
Keywords: delta-9-tetrahydrocannabinol; THC; Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- delta-9-tetrahydrocannabinol (Active Comparator): Subjects will be randomized to receive 3 doses Namisol® (3 mg, 5 mg, 6,5 mg)
  Interventions: Drug: delta-9-tetrahydrocannabinol
- Placebo (Placebo Comparator): The control product is placebo, consisting of a tablet with similar appearance and taste of the test product.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: delta-9-tetrahydrocannabinol — During the intervention phases, subjects will be randomly allocated to receive 1 of 3 doses Namisol®: 3 mg, 5 mg, 6,5 mg (or placebo) The washout period between the intervention periods will be at least 2 weeks.
  Other Names: Namisol; Cannabis; ECP002A
  Arms: delta-9-tetrahydrocannabinol
Drug: Placebo — On each intervention day the subjects will receive the same amount of drugs in order to insure the blinding of the study
  Other Names: The control product is placebo
  Arms: Placebo

SUMMARY:
The results of phase I Namisol® study (Klumpers et al. Br J Clin Pharmacol, 2012), implicate that Namisol® may have a favorable PK and PD characteristics and is safe to use in people. However, the study included only young adults with a mean age of 21.4 years. In a previous THC study, subjects age has been associated with treatment response and tolerance of adverse reactions. This association was not supported by Lane et al. and Volicer et al.

There is concern about the safety and tolerability of THC in the elderly population. This is because, elderly persons in general have higher risk of adverse drug reactions due to a combination of physiological factors such as decreasing in lean body mass, the reduction of renal and hepatic clearance, and medical comorbidity which can lead to polypharmacy and drug-drug interactions. Therefore, data from the phase I trial cannot be translated directly to an elderly (and likely more vulnerable) population. This makes it important to evaluate the safety and tolerability profiles of different Namisol® doses in the elderly. In our study in progress "Delta-THC in Behavioral Disturbances in Dementia", the Namisol® doses of 0,75 mg and 1,5 mg are, until now, well tolerated by elderly subjects. These doses are, however, very low in comparison with the doses used in phase I study with young adults (5 mg, 6,5 mg and 8 mg). The current study on the safety and tolerability of relatively high doses of Namisol® will help us in the future to provide broad advice on the therapeutic index and safety profile of Namisol® in the elderly population.

DETAILED DESCRIPTION:
Subjects will visit the site 5 times. The first visit, is a 2 hour screening visit for eligibility in which volunteers after signing informed consent will have a medical history, physical examination, ECG, hematological and biochemical blood tests, Mini Mental State Examination (MMSE), Geriatric Depression scale (GDS-30) and body sway test.

Eligible subjects will be randomly allocated to receive three doses Namisol® (3 mg or 5 mg or 6,5 mg) and placebo in double-blind crossover design (visit 1 to 4). The wash-out period between visits will be at least 2 weeks to a maximum of 4 weeks. Each visit will be preceded by baseline assessment measures. The safety and tolerability profiles of Namisol® will be evaluated on each intervention visit by using a standardized THC adverse effects checklist and self-reporting, vital signs, 12-lead ECG, body sway, Visual Analogue Scales (subtest feeling high), and Test for Attentional Performance (TAP, subtest alertness) and a follow up phone call the following day. Four blood samples will be collected on each visit to determine the relationship between the pharmacodynamic effects (VAS-feeling high, TAP-alertness and body sway) and the plasma concentrations of THC and its active metabolites 11-OH-THC and THC-COOH. In addition, a blood sample will be only collected on the first intervention day for genotyping of cytochrome P450 enzymes CYP2C9 CYP2C19 and CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy old person as established by medical history, physical examination, electrocardiography, results of hematological and biochemical blood tests on screening.
* Age 65 years
* Body mass index between 18.0 and 30 kg m-2
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations

Exclusion Criteria:

* Regular cannabis user, defined as: smoking one or more joints per week
* Documented history of sensitivity/idiosyncrasy to cannabis
* Relevant history or presence of severe pulmonary disorders [e.g. COPD GOLD III or IV], serious cardiovascular disorders [e.g. myocardial infarction < 6 months ago; atrial fibrillation; heart failure NYHA III or IV; severe heart valve disease, orthostatic hypotension defined as systolic drop of 20 mm Hg Safety and Tolerability of Namisol in the Elderly Page 8 Version 2, 10 07 2012 or diastolic drop of 10 mm Hg], seizures, migraine, psychiatric disorders [e.g. depression (based on documented history or GDS-30 on screening ≥ 10); mania; psychosis; dementia], cognitive impairment [based on documented history or MMSE on screening < 28, significant renal (GFR < 30 ml/min) or hepatic disorders [e.g. cancer, cirrhosis. ALT or AST ≥ twice the upper limit of normal], diabetes mellitus, coagulation disorders
* Inability to understand the nature and extent of the trial and the procedures required
* Current alcohol abuse or use of more than 2 alcoholic consumptions daily
* History of, or current drug abuse
* Using drugs that are inhibitors of CYP2C9, CYP2C19 and CYP3A4 (see appendix 13.3)
* Participation in a drug trial within 60 days prior to the first intervention day
* Donation of blood within 60 days prior to the first intervention day
* Known lactose intolerance
* Using more than six units of (methyl)xanthine products per day (e.g. coffee, tea, cola, chocolate)
* Smoking more than ten cigarettes per day
* High fall-risk (based on body sway test)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
THC adverse effects checklist and self-reporting by the subjects | Pre dose, 0h30m, 1h30m and at 2h30m post ingestion
  Safety and tolerability of Namisol® will be evaluated by assessing the incidence and severity of adverse events on each intervention visit by using a standardized THC adverse effects checklist and self-reporting by the subjects.

SECONDARY OUTCOMES:
Body Sway Test (SwayStar™) | Pre dose, 0h40m, 0h55m and at 2 hour post ingestion
  On each intervention visit the body sway will be assessed by using the SwayStar®.The SwayStar® device consists of 2 digitally-based angular velocity transducers and is worn on the lower back (at the level of the lumbar spine, lumbar 2-3). It is a wireless device, which makes it possible to examine subjects" balance while walking. The transducers can accurately assess angular movement and angular velocities in 2 directions: anterior-posterior (pitch plane) and mediolateral (roll plane)
Visual analogue scales, subtest "feeling high" | Pre dose, 0h40m, 0h55m and at 2 hour post ingestion
  The Bowdle visual analogue scales (VAS) of psychedelic effects will be performed on each intervention visit in order to measure subjective feeling high
Test for Attentional Performance (TAP), subtest alertness | Pre dose, 0h40m, 0h55m and at 2 hour post ingestion
  On each intervention visit the alertness of subjects will be measured by using the TAP. The TAP subtest "Alertness" measures the subject's ability to respond to a visual stimulus and to increase the attentional level in expectance of a stimulus of high priority. The computer-assisted test is given under 2 conditions: (1) Simple reaction time to a visual stimulus (Greek cross) appearing at randomly varying intervals on the monitor screen is measured. (2) In the second condition, the visual stimulus (= critical stimulus) is preceded by a cue sound presented as warning tone.
Plasma concentrations of THC and its active metabolites 11-OH-THC and THC-COOH | Pre dose, 0h40m, 0h55m and at 2 hour post ingestion
  Four blood samples will be collected on each visit to determine the relationship between the pharmacodynamic effects ( using VAS-feeling high, TAP-alertness and body sway) and the plasma concentrations of THC and its active metabolite 11-OH-THC and THC-COOH.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Olde Rikkert, prof. dr., Principal Investigator — Radboud University Medical Center Nijmegen
Locations (1):
- Radboud University Medical Centre, department of Geriatrics, Nijmegen, Gelderland, Netherlands